CLINICAL TRIAL: NCT00964847
Title: Lifestyle Modification and Blood Pressure Study
Acronym: LIMBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01AT004921-01A1 (NIH)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: High Blood Pressure
Keywords: hypertension; cardiovascular disease; yoga
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Blood pressure education/walking program (Active Comparator)
  Interventions: Behavioral: Blood pressure education/walking program
- Combined intervention (Active Comparator)
  Interventions: Behavioral: Yoga exercise program; Behavioral: Blood pressure education/walking program
- Yoga Exercise Program (Experimental)
  Interventions: Behavioral: Yoga exercise program

INTERVENTIONS:
Behavioral: Yoga exercise program — Subjects in the yoga exercise program participate in structured bi-weekly 1.5 hour yoga classes held at a yoga studio as well as develop a weekly hour-long home practice over the 6 months of the study.
  Other Names: YP
  Arms: Combined intervention; Yoga Exercise Program
Behavioral: Blood pressure education/walking program — The program will consist of small group health education classes and a walking program. Subjects will be expected to attend a dietician-led nutrition class twice a month. On alternate weeks the subjects will be given either motivational talks about a variety of topics including weight loss, walking programs, and healthy lifestyle choices or they will be given educational DVDs or literature to read on the weeks that they are not attending a BPEP class. These subjects will all receive 12 nutrition classes and 12 motivational experiences. The subjects will also be expected to walk 6 days a week gradually increasing to 180 minutes of walking per week or 10,000 steps per day.
  Other Names: BPEP
  Arms: Blood pressure education/walking program; Combined intervention

SUMMARY:
The purpose of this study is to compare the effects of 24 weeks of either a blood pressure education and walking program versus a yoga exercise program versus the combined intervention of blood pressure education and yoga on reducing mild to moderate high blood pressure in pre-hypertension and stage 1 hypertension subjects.

DETAILED DESCRIPTION:
The study is a non-blinded, randomized controlled trial to assess the safety and efficacy of 24 weeks of a structured yoga exercise program (YP) versus a blood pressure education and walking program (BPEP) versus the combined intervention on reducing mild to moderate high blood pressure in adults with pre-hypertension or stage 1 hypertension. This will be done through a single center trial using a parallel design. All potential subjects will be screened first by telephone and then by 2 outpatient visits at the Clinical and Translational Research Center (CTRC) at the hospital of the University of Pennsylvania. Eligible subjects will then make 3 visits to the CTRC where they will be admitted overnight to have non-invasive 24-hour recordings of BP, as well as have periodic blood, urine and saliva collections. The entire study duration is 28 weeks (24 weeks post-randomization) and includes a total of 7 evaluation visits (including 2 functional magnetic resonance imaging visits) and a termination visit. Subjects will be randomized to YP, BPEP or the combined intervention of YP and BPEP.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to give written informed consent.
* Age > 18 years, but < 75 years.
* BP criteria: Systolic Blood Pressure (SBP) of > 130, but < 160 mm Hg.
* Willing to comply with all study-related procedures.

Exclusion Criteria:

* Subjects who are pregnant or post partum < 3 months.
* Subjects currently taking BP lowering medications or dietary supplements (magnesium, potassium, calcium > 1200 mg/day, fish oils, ephedra, hawthorn, forskolin, etc…).
* Stage II HTN (SBP > 160 mmHg OR diastolic blood pressure (DBP) > 100 mmHg).
* Non-dominant arm circumference > 50 cm.
* BMI > 40.0 kg/m2.
* Practicing yoga >1x/month in the previous 6 months.
* Received/used experimental drug or device within 30 days prior to screening, or donated blood > 1 pint within 8 weeks of screening.
* Diabetes mellitis.
* Established cardiovascular disease.
* Known arrhythmias or cardiac pacemakers.
* Current users (within 30 days) of any tobacco products.
* History of renal insufficiency (glomerular filtration rate < 60 ml/min).
* Women consuming > 7 alcoholic drinks/week; men consuming > 14 drinks/week.
* Known autonomic neuropathy.
* Known secondary cause of HTN (renal artery stenosis, pheochromocytoma, coarctation of aorta, hyperaldosteronism).
* Benzodiazepine, anti-psychotic drugs (3 month stable use of SSRIs are allowed), or steroid use.
* Known severe musculoskeletal problems such as spinal stenosis that may limit participation in yoga.
* Use of other mind/ body therapies such as Qi Gong, Tai Chi, meditation.
* Lack Internet access.
* Presence of non-removable metallic foreign object, surgically implanted electrical device, surgically placed metallic clip (aneurysm clip), ear implants, any history of metal implants in the eye.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2009-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory blood pressure | baseline, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Cerebral blood flow | baseline, 12 weeks, 24 weeks
Urinary Isoprostane | baseline, 12 weeks, 24 weeks
serum asymmetric dimethylarginine (ADMA) | baseline, 12 weeks, 24 weeks
salivary cortisol | baseline, 12 weeks, 24 weeks
psychological measures of mood, perceived stress and health competence | baseline, 12 weeks, 24 weeks
physiological measures of flexibility | baseline, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Cohen, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital at the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cohen D, Townsend RR. Yoga and hypertension. J Clin Hypertens (Greenwich). 2007 Oct;9(10):800-1. doi: 10.1111/j.1751-7176.2007.tb00008.x. No abstract available. PMID 17917509
- [Background] Cohen DL, Wintering N, Tolles V, Townsend RR, Farrar JT, Galantino ML, Newberg AB. Cerebral blood flow effects of yoga training: preliminary evaluation of 4 cases. J Altern Complement Med. 2009 Jan;15(1):9-14. doi: 10.1089/acm.2008.0008. PMID 19769471
- [Background] Cohen DL, Bloedon LT, Rothman RL, Farrar JT, Galantino ML, Volger S, Mayor C, Szapary PO, Townsend RR. Iyengar Yoga versus Enhanced Usual Care on Blood Pressure in Patients with Prehypertension to Stage I Hypertension: a Randomized Controlled Trial. Evid Based Complement Alternat Med. 2011;2011:546428. doi: 10.1093/ecam/nep130. Epub 2011 Feb 14. PMID 19734256
- [Derived] Cohen DL, Boudhar S, Bowler A, Townsend RR. Blood Pressure Effects of Yoga, Alone or in Combination With Lifestyle Measures: Results of the Lifestyle Modification and Blood Pressure Study (LIMBS). J Clin Hypertens (Greenwich). 2016 Aug;18(8):809-16. doi: 10.1111/jch.12772. Epub 2016 Jan 15. PMID 26773737
- [Derived] Cohen DL, Bowler A, Fisher SA, Norris A, Newberg A, Rao H, Bhavsar R, Detre JA, Tenhave T, Townsend RR. Lifestyle Modification in Blood Pressure Study II (LIMBS): study protocol of a randomized controlled trial assessing the efficacy of a 24 week structured yoga program versus lifestyle modification on blood pressure reduction. Contemp Clin Trials. 2013 Sep;36(1):32-40. doi: 10.1016/j.cct.2013.05.010. Epub 2013 May 27. PMID 23721984